CLINICAL TRIAL: NCT04227236
Title: Interventions to Improve Reproductive Health Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: dfusion Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R41HD094406 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2020-01-13 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Teacher Training
Keywords: Sexual; health
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two groups: in-person training or e-based virtual training.
Masking Description: No masking was done as the assignment was evident based on the type of training offered. However, participants were unaware of the other options.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-based virtual training (Experimental): Participants in the e-based virtual training (up to 8 participants per session) will be placed at one of eight computers (with headphones), which we estimate will take less time (about 40 minutes), due to the individualized learning and 1:1 nature of the training instead of 1:15. Participants will complete the condom-line up facilitator training module that corresponds to the Making Proud Choices curriculum.
  Interventions: Other: E-based virtual facilitator training for Making Proud Choices
- In-person training (Active Comparator): Participants in-person training will participate in a class with 15-20 participants like the usual MPC training environment. The training will last 1 hour. Like the e-based virtual training, participants will complete the condom-line up facilitator training module that corresponds to the Making Proud Choices curriculum.
  Interventions: Other: In-person facilitator training for Making Proud Choices

INTERVENTIONS:
Other: E-based virtual facilitator training for Making Proud Choices — Participants complete the Making Proud Choices (MPC) facilitator training using an e-based virtual trainer on a computer. Making Proud Choices! (MPC) is an evidence-based pregnancy and HIV/STI risk-reduction program for youth. The facilitator training prepares educators to effectively deliver the MPC curriculum.
  Arms: E-based virtual training
Other: In-person facilitator training for Making Proud Choices — Participants complete the Making Proud Choices (MPC) facilitator training using the standard in-person training method. Making Proud Choices! (MPC) is an evidence-based pregnancy and HIV/STI risk-reduction program for youth. The facilitator training prepares educators to effectively deliver the MPC curriculum.
  Arms: In-person training

SUMMARY:
The proposed virtual training prototype will provide Making Proud Choices (MPC) facilitator trainees the opportunity to make decisions, build facilitator skills, practice core concepts and enhance self-efficacy with a virtual audience programmed to display a range of behaviors and emotions, simulating a true-to-life experience with immediate feedback. Seventy-two adults who have experience working with adolescents but not with MPC, STI, or pregnancy prevention education will receive MPC training. Participants will be randomly assigned to either: 1) virtual training in the MPC module on condom use n=36), or 2) dfusion/ETR's traditional in-person training in the same module (n=36). Using mixed methods (survey, focus groups, observations), the project will evaluate the virtual training's impact on STI/pregnancy prevention knowledge, teaching efficacy, and teaching skills and its usability, feasibility, and acceptability.

DETAILED DESCRIPTION:
Dfusion, in partnership with the RAND Corporation, Allen Interactions and Dr. Loretta Jemmott (MPC developer), proposes to develop an online avatar-based virtual training that can make MPC training more accessible while still being as effective as in-person. In this Phase I STTR, we will develop and test a prototype of the online, avatar-based virtual training for activities of MPC and test it with 72 adults who have experience working with adolescents (but not with MPC or any HIV/STI/teen pregnancy risk-reduction program). At random, 36 will receive traditional in-person MPC training, and 36 will receive avatar-based MPC training. The avatar group (n=36) will be compared to the in-person group (n=36) on their STI/pregnancy prevention knowledge, teaching efficacy, and teaching skills.

The scientific premise is that avatar-based virtual training will prepare educators to implement the popular evidence-based MPC as effectively as traditional (and expensive) face-to-face trainings. The specific aims are:

* Aim 1: Develop a prototype for a novel, online avatar-based virtual training for select components of the evidence-based STI/pregnancy risk reduction program Making Proud Choices.
* Aim 2: Using mixed methods (survey, focus groups, observations), evaluate the avatar-based training's preliminary impact on facilitator STI/pregnancy prevention knowledge, teaching efficacy, and teaching skills compared to in-person training, as well as its usability and acceptability.

By developing novel tools/platforms to improve the dissemination and implementation of evidence-based behavioral interventions to prevent STIs/teen pregnancy, this application is in line with the priorities of the NICHD Population Dynamics Branch, which supports reproductive health research on STIs and family planning. If successful, not only will dfusion proceed to Phase II, but the findings could inform other nascent efforts to develop avatar facilitator trainings that could make a range of evidence-based programs more accessible to community-based organizations.

ELIGIBILITY:
Inclusion Criteria:

* age 21+ and have no prior experience with MPC or providing STI or pregnancy prevention education

Exclusion Criteria:

* non-English speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dfusion, Inc, Scotts Valley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the raw data files and codebooks available for public use within one year of the final year of funding. We will make the dataset and associated documentation available outside our team under a data-sharing agreement that provides for (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology and (3) a commitment to destroying or returning the data after analyses are completed. Identifiers will never be included in these shared files. Individual researchers can contact the PIs for data and through filling out a data request and use form that we will create for the purposes of data sharing. Researchers can access the data through RAND's restricted-access server with password protection after their request is reviewed and approved by our institution officials.
Supporting Information: SAP, CSR
Time Frame: We will make the data and supporting information available within one year of the final year of funding of the project. No end date is determined.
Access Criteria: Individual researchers can contact the PIs for data and through filling out a data request and use form that we will create for the purposes of data sharing. Researchers can access the data through RAND's restricted-access server with password protection after their request is reviewed and approved by our institution officials.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-based Virtual Training | In-person Training
Started | 31 | 22
Completed | 31 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-based Virtual Training | In-person Training | Total
Number analyzed (Participants) | 31 | 22 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (13.4) | 40.8 (14.1) | 38.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 13 | 11 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity: Hispanic | 3 | 4 | 7
  Race and ethnicity: Non-Hispanic White | 17 | 11 | 28
  Race and ethnicity: Non-Hispanic Black | 4 | 2 | 6
  Race and ethnicity: Non-Hispanic Asian | 6 | 2 | 8
  Race and ethnicity: Multiple Race | 1 | 2 | 3
  Race and ethnicity: unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 22 | 53

OUTCOME MEASURES:

1. Primary Outcome: Implementation Fidelity: Conducting Condom Line-up
Description: Participants teach an activity that is video recorded and coded for fidelity to the Making Proud Choices curriculum. Participants are scored on the completion of multiple curriculum tasks by two coders as 2=done correctly, 1=done partially correct, or 0=not done correctly. This particular measure was a single item about the degree to which the teacher correctly conducted the condom line up activity.
Time Frame: up to 1 hour post teacher training
Measure: Mean (Standard Deviation); unit: score on an item
Groups:
- E-based Virtual Training: Participants in the e-based virtual training (up to 8 participants per session) were placed at one of eight computers (with headphones), which took about 40 minutes. Participants completed the condom-line up facilitator training module that corresponds to the Making Proud Choices curriculum. Participants completed the Making Proud Choices (MPC) facilitator training using an e-based virtual trainer on a computer. Making Proud Choices! (MPC) is an evidence-based pregnancy and HIV/STI risk-reduction program for youth. The facilitator training prepares educators to effectively deliver the MPC curriculum.
- In-person Training: Participants in-person training participated in a class with 15-20 participants like the usual MPC training environment. The training lasted 1 hour. Like the e-based virtual training, participants completed the condom-line up facilitator training module that corresponds to the Making Proud Choices curriculum. Participants completed the Making Proud Choices (MPC) facilitator training using the standard in-person training method. Making Proud Choices! (MPC) is an evidence-based pregnancy and HIV/STI risk-reduction program for youth. The facilitator training prepares educators to effectively deliver the MPC curriculum.
Arm/Group | E-based Virtual Training | In-person Training
Number analyzed (Participants) | 31 | 22
score on an item | 1.67 (0.44) | 1.26 (0.56)

2. Primary Outcome: Training Knowledge of Condom Line-Up Activity
Description: 7-item survey measure of knowledge related to condom safety and objectives of the condom line-up module of Making Proud Choices. Responses were coded as correct (1) and incorrect (0). Averaging together the 0s and 1, we calculated a percentage correct for the whole 7 item survey, with 100% being all correct, and 0% being all incorrect.
Time Frame: 30 minutes before teacher training and 30 minutes after training
Population: Total population separated by e-based and in-person training
Measure: Mean (Standard Deviation); unit: Percent correct
Arm/Group | E-based Virtual Training | In-person Training
Number analyzed (Participants) | 31 | 22
Percent correct
  Pre-training | 63.3 (21.1) | 66.7 (19.3)
  Post-training | 96.6 (4.5) | 100.0 (0.0)

3. Primary Outcome: Change in Teaching Self-efficacy
Description: 4-item self-efficacy measure assessing confidence in teaching condom safety, rated from 1 (not at all) to 7(extremely). Scores were averaged to create a self-efficacy scale score. Change scores were calculated by subtracting scores Post-Pre Training.
Time Frame: 30 minutes before teacher training and 30 minutes after training
Population: in-person and online training participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-based Virtual Training | In-person Training
Number analyzed (Participants) | 31 | 22
score on a scale | .59 (.99) | .75 (.69)

4. Primary Outcome: Implementation Fidelity: Discuss Steps in Condom Use
Description: Participants teach an activity that is video recorded and coded for fidelity to the Making Proud Choices curriculum. Participants are scored on the completion of multiple curriculum tasks by two coders as 2=done correctly, 1=done partially correct, or 0=not done correctly. This particular measure was a single item about the degree to which the teacher correctly discussed the steps in the activity on how to use a condom properly.
Time Frame: 1 hour after training
Measure: Mean (Standard Deviation); unit: score on an item
Arm/Group | E-based Virtual Training | In-person Training
Number analyzed (Participants) | 31 | 22
score on an item | 1.15 (0.88) | 0.79 (0.93)

5. Secondary Outcome: Acceptability of Training
Description: 19-item measure of perceived acceptability of Making Proud Choices e-based facilitator training. The overall score, which is an average of all 19 items, uses a 7-point scale (strongly agree to strongly disagree). Higher scores equal greater acceptability. Thus, the high score is 7 (training perceived as most acceptable). The low score is 1 (training perceived as the least acceptable).
  Only the participants of the E-based Virtual Training group were asked these questions.
Time Frame: 30 minutes after teacher training
Population: Only the participants of the E-based Virtual Training were asked these questions because they only applied to the online training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-based Virtual Training
Number analyzed (Participants) | 31
score on a scale | 5.80 (1.12)

6. Secondary Outcome: Applicability of Training
Description: 10-item measure of perceived applicability of Making Proud Choices e-based facilitator training. Items were rated on a 7-point scale (strongly agree to strongly disagree). All items were averaged together to create a total score, with higher scores representing greater perceptions of applicability. Thus, the high score is 7 (training perceived as most applicable). The low score is 1 (training perceived as the least applicable).
  Only participants in the E-based Virtual Training group were asked these questions.
Time Frame: 30 minutes after teacher training
Population: Only participants in the E-based Virtual Training group were asked these questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-based Virtual Training
Number analyzed (Participants) | 31
score on a scale | 5.55 (1.18)

7. Secondary Outcome: Overall Impression
Description: Participants overall impressions of the training were assessed using 4 item measure, rated on a 7-point Likert scale ("very difficult to use" to "very easy to use", "very boring" to "very interesting", "very amateurish" to "very professional", and "very basic" to "very informative"). Items were average to create an overall impression score, with higher scores reflecting greater overall impression. Thus, the high score is 7 (training perceived with the highest favorable impression). The low score is 1 (training perceived with the least favorable impression).
  Only participants of the E-based Virtual Training group answered these questions.
Time Frame: 30 minutes after teacher training
Population: Only participants of the E-based Virtual Training group answered these questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-based Virtual Training
Number analyzed (Participants) | 31
score on a scale | 5.46 (1.15)

ADVERSE EVENTS:
Time Frame: 1 day (day of the training)
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, does NOT differ from the clinicaltrials.gov definitions.
Arm/Group | E-based Virtual Training | In-person Training
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/22
Other Adverse Events (participants affected / at risk) | 0/31 | 0/22

LIMITATIONS AND CAVEATS:
Our findings are limited by a small sample size, which is typical for a Phase I SBIR grant meant to be a "proof of concept" study. Recruitment included adults (18 years or older) with interest in the study and no prior experience with MPC rather than teachers or community-based youth leaders who are likely the target audience for this training.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT04227236/Prot_SAP_ICF_000.pdf